CLINICAL TRIAL: NCT03148301
Title: Spina Bifida in Daily Life: an Exploratory Study
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S60433
Record Dates: First submitted 2017-05-08; First posted 2017-05-10 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Spina Bifida
MeSH Terms: conditions — Spinal Dysraphism | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Spina Bifida: Adults with and parents of children with Spina Bifida followed by the team in UZ Leuven will be asked to complete a survey
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — Survey

SUMMARY:
Spina Bifida can lead to physical neurocognitive and psychological symptoms. Still little is know about the daily impact of spina bifida on participation possibilities in social life. This exploratory research project want to investigate which lif choices patients with spina bifida has to make and in which way their daily life is organized. In a second part, quality of life will be measured and we hope to discover some dynamics in order to improve patient care.

DETAILED DESCRIPTION:
This exploratory research project wants to investigate how patients with spina bifida live their daily life and which impact spina bifida has on their choices of life. This will be done by a survey that will ask questions about different domains in life: demographic variables, education, work, social functioning, spare time, housing, mobility, independency and quality of life. The survey is based on empirical findings in literature. The quality of life questioning is based on the SF36. The survey will be done once during a clinical consultation.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Spina Bifida

Exclusion Criteria:

* Not able to read or write Dutch

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Spina Bifidat patients that are seen on the consultation or day care unit of UZ Leuven
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Descriptive statistics about life choices | 1 year
  Descriptive statistics about life choices measured by the answers of the survey of Spina Bifida patients

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No